CLINICAL TRIAL: NCT04530734
Title: Blood Concentration in Lorazepam and Treatment in Adult Catatonia
Acronym: PHARMAPREDICAT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_17; 2019-A01208-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-06-25; First posted 2020-08-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Catatonia
MeSH Terms: conditions — Catatonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Catatonia is a severe form of psychomotor disturbance with a heterogenous presentation. It affects approximately 10% of acute psychiatric inpatients. According to the fifth edition of DSM-5 the diagnosis of catatonia can be made when three or more symptoms from the twelve following are present : catalepsy, waxy flexibility, stupor, agitation, mutism, negativism, posturing, mannerisms, stereotypies, grimacing, echolalia, echopraxia. It can occur in various psychiatric diseases, including mood disorders or schizophrenia, but also in various non-psychiatric disorders [metabolic disturbances, viral infections (including HIV), typhoid fever, heat stroke, and autoimmune disease].

Benzodiazepines, especially LORAZEPAM, are the most common initial treatment, with a remission rate of approximately 70-80 %, regardless of the cause or the clinical manifestations. This first line treatment is titrated gradually according to the therapeutic response over a few days up to 20-25 mg per day. Electroconvulsive therapy (ECT) is initiated on patients with catatonia who do not respond to benzodiazepines.

Interestingly, pharmacogenetic variants can alter the metabolism of lorazepam (e.g., the UGT2B15 * 2 allele slows it down).

The main objective of this study is to assess the link between clinical response to lorazepam, residual plasma concentrations of lorazepam after 72 hours of fixed dosage, and the existence of genetic polymorphisms modifying the metabolism of lorazepam. Our hypothesis is that non-responding patients have lowered blood concentrations of lorazepam associated to a genetic profile of rapid metabolism. Evaluating the predictive factors of the response to treatment would allow early and precise identification of non-responder patients in order to adapt their first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* catatonia according DSM-5

Exclusion Criteria:

* Subject is less than 18 years of age
* Subject is pregnant at the time of the study
* Subject/legal guardian unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 102 patients with catatonia. 70 responder patients, 32 non responder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of lorazepam measured after 72 hours of treatment with lorazepam at fixed dose | at 72 hours of treatment with lorazepam
  Compare the residual plasma concentration of lorazepam after 72 hours of taking fixed-dose lorazepam between responder and non-responder patients defined by the persistence of this diagnosis despite a daily dosage of 24 mg of lorazepam for 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ali AMAD, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Fontan, CHU lille, Lille, France